CLINICAL TRIAL: NCT00597662
Title: Safety Study of Polylactide-Caprolactone-Trimethylenecarbonate Copolymer for Post-Operative Adhesion Prophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Dr. D. Wallwiener, Universitäts-Frauenklinik Tübingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SUP-002
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Device: polylactide-caprolactone-trimethylenecarbonate copolymer
- 2 (Active Comparator)
  Interventions: Device: Icodextrin 4%

INTERVENTIONS:
Device: polylactide-caprolactone-trimethylenecarbonate copolymer — Polylactide-caprolactone-trimethylenecarbonate copolymer membrane is applied directly over the surgical scar on the visceral peritoneum
  Arms: 1
Device: Icodextrin 4% — 1 liter icodextrin 4% is instilled into the peritoneal cavity at the end of the operation
  Arms: 2

SUMMARY:
The purpose of this study is to compare adhesion prophylaxis with polylactide-caprolactone-trimethylenecarbonate copolymer to icodextrin 4% in terms of safety, side effects and usability in addition to gaining early evidence of the effectiveness of polylactide-caprolactone-trimethylenecarbonate copolymer.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* sex female
* laparoscopic myomectomy indicated
* ability and intention to conform to the study protocol
* written informed consent

Exclusion Criteria:

* pregnancy
* indication for laparotomy
* inflammatory bowel disease
* additional surgical interventions
* known or suspected intollerance or hypersensibility to the interventions
* chronic pain
* systemic corticoids or irradiation
* alcohol abuse or other substance abuse
* clinical signs of malignancy
* psychiatric or neurological disease
* participation in another clinical trial within 30 days
* inability to understand the purpose of the trial or to conform to the study protocol
* absence of written informed consent
* inflammation of pelvic organs
* presence of adhesions which lead to a conversion from laparoscopy to laparotomy
* concurrent therapy with corticoids, anti-neoplastic agents or irradiation
* maintenance therapy with non-steroidal anti-inflammatory drugs or analgesics

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Difference in visual analogue pain score on visit 8 after discharge minus visit 1 on admission | 3 months

SECONDARY OUTCOMES:
Use of analgesia | 1, 2 and 3 days
Post-operative pyrexia | 3 months
Post-operative infection | 3 months
Requirement for re-operation | 3 months
Dysmenorrhoea | 3 months
Dyspareunia | 3 months
Constipation | 3 months
Diarrhoea | 3 months
Nausea | 3 months
Duration of adhesion prophylaxis | Day 1
Usability as assessed by surgeon | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Prof. Dr., Study Chair — Universitäts-Frauenklinik Tübingen
Locations (1):
- Universitäts-Frauenklinik Tübingen, Tübingen, Baden-Wurttemberg, Germany